CLINICAL TRIAL: NCT00037635
Title: A Phase 3 Study to Assess the Efficacy and Safety of an Oral Calcimimetic Agent (AMG 073) in Secondary Hyperparathyroidism of End Stage Renal Disease Treated With Hemodialysis
Brief Title: A Study of an Investigational Medication for the Treatment of Secondary Hyperparathyroidism in Dialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20000172
Record Dates: First submitted 2002-05-17; First posted 2002-05-20 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Secondary Hyperparathyroidism; End Stage Renal Disease
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Kidney Failure, Chronic | interventions — Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- AMG 073 (Experimental)
  Interventions: Drug: AMG 073
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 073 — 30 mg QD orally 60 mg QD orally 90 mg QD orally 120 mg QD orally 180 mg QD orally
  Arms: AMG 073
Drug: Placebo — 30 mg QD orally 60 mg QD orally 90 mg QD orally 120 mg QD orally 180 mg QD orally
  Arms: placebo

SUMMARY:
This 6 month long study will assess an investigational medication for patients on dialysis with secondary hyperparathyroidism. The study will look at the effects on parathyroid hormone, calcium and phosphorus levels.

ELIGIBILITY:
* Patients must be receiving hemodialysis; * Have elevated parathyroid hormone levels; * Not be pregnant or nursing; and * Not have had a heart attack in the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2001-12; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of AMG 073 compared with placebo by determining the proportion of subjects with a mean intact parathyroid hormone (iPTH) value <= 250 pg/mL (26.5 pmol/L) during the efficacy assessment phase. | efficacy assessment phase (last 14 weeks of treatment)

SECONDARY OUTCOMES:
To evaluate the efficacy of AMG 073 compared with placebo by determining: percentage change from baseline in mean calcium x phosphorus product (Ca x P) during the efficacy assessment phase | efficacy assessment phase (last 14 weeks of treatment)
To evaluate the efficacy of AMG 073 compared with placebo by determining: changes in self-reported cognitive function from baseline to the end of the efficacy assessment phase | efficacy assessment phase (last 14 weeks of treatment)
To evaluate the safety of AMG 073 compared with placebo. | entire study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Martin KJ, Juppner H, Sherrard DJ, Goodman WG, Kaplan MR, Nassar G, Campbell P, Curzi M, Charytan C, McCary LC, Guo MD, Turner SA, Bushinsky DA. First- and second-generation immunometric PTH assays during treatment of hyperparathyroidism with cinacalcet HCl. Kidney Int. 2005 Sep;68(3):1236-43. doi: 10.1111/j.1523-1755.2005.00517.x. PMID 16105056
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com